CLINICAL TRIAL: NCT05702853
Title: A Phase 1b Dose Escalation Study of Metabolically Fit CD19 Chimeric Antigen Receptor (CAR) T Cells With CD34 Selection Markers in Adult Patients With Relapsed or Refractory CD19 B-Cell Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Metabolically Fit CD19 CAR T-cell Therapy With CD34 Selection in Patients With CD19+ Relapsed/Refractory NHL, CLL/SLL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 103351
Record Dates: First submitted 2022-12-07; First posted 2023-01-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: B-cell Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: NHL; CLL; SLL; CD19; CAR-T; CD34
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1 (Experimental): 1 x 10^6 transduced T cells/kg (± 20%)
  Interventions: Drug: Cyclophosphamide injection; Drug: Fludarabine Injection; Biological: CD19-CD34t metabolically programmed CAR transduced T-cells
- Dose Level 2 (Experimental): 1.5 x 10^6 transduced T cells/kg (± 20%)
  Interventions: Drug: Cyclophosphamide injection; Drug: Fludarabine Injection; Biological: CD19-CD34t metabolically programmed CAR transduced T-cells
- Dose Level 3 (Experimental): 2 x 10^6 transduced T cells/kg (± 20%)
  Interventions: Drug: Cyclophosphamide injection; Drug: Fludarabine Injection; Biological: CD19-CD34t metabolically programmed CAR transduced T-cells

INTERVENTIONS:
Drug: Cyclophosphamide injection — 500 mg/m2 IV over 30-60 minutes +/- 10 minutes before Fludarabine Days -5, -4, - 3
Drug: Fludarabine Injection — 30 mg/m2 IV over 30-60 minutes +/- 10 minutes after cyclo- phosphamide infusion Days -5, 4, -3
Biological: CD19-CD34t metabolically programmed CAR transduced T-cells — Cells are to be infused intravenously (IV) over 30 minutes or less via nonfiltered tubing either by gravity or a peristaltic pump, gently agitating the bag during infusion to prevent cell clumping

SUMMARY:
This is a single-center, nonrandomized, open-label dose-escalation study followed by dose-expansion of CD19- CD34t metabolically programmed CAR T-cell therapy in adult patients with relapsed or refractory CD19 B-cell non-Hodgkin lymphoma (NHL) or chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
Although CD19 CAR T-cell therapy is a dynamic scientific and clinical breakthrough for CD19+ NHL, issues still remain in terms of relapse, toxicity, and availability. This trial will incorporate a CD34 tag (CD34t) into the CAR T-cell construct, thus allowing a more purified CAR T-cell product via CD34 selection. This purification step will hopefully lead to an improvement in safety/toxicity. Furthermore, the issue of CD19 CAR T-cell relapse has been linked to a lack of CAR T-cell fitness. With the knowledge that Th1 T-cell subsets have improved effector function and Th17 T-cell subsets have improved persistence, the investigators plan to expose the collected T-cells to priming conditions that lead to a metabolically enhanced CAR-T cell product akin to a Th1/17 hybrid cell. The investigators hypothesize that these metabolically programmed CD19 CAR-T cells will yield a high- quality product with enhanced persistence and anti-tumor efficacy when purified based on CD34t expression.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for study participation must meet all of the following criteria:

1. Disease Related Criteria

   Participants must have histologic confirmation of one of the following:
   1. CD19+ aggressive non-Hodgkin lymphoma including any of the following subtypes

      * Diffuse Large B-cell Lymphoma, not otherwise specified
      * DLBCL, germinal-center B-cell type (GCB)
      * DLBCL, activated B-cell type (ABC)
      * T-cell histiocyte-rich B-cell lymphomas (THRBCL)
      * Primary cutaneous DLBCL, leg type
      * Intravascular large B cell lymphoma
      * EBV+ DLBCL, NOS
      * DLBCL associated with chronic inflammation
      * HHV8+ DLBCL, NOS
      * High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement(double hit lymphoma)
      * High grade B-cell lymphoma, NOS
      * Primary mediastinal B-cell lymphoma
      * B-cell Lymphoma, unclassifiable with features intermediate between DLBCL and Hodgkin lymphoma, as well as with features intermediate between DLBCL and Burkitt lymphoma
      * Follicular lymphoma grade 3B
      * Transformation of indolent lymphoma (i.e. CLL, MZL, FL, Waldenstrom's lymphoma,etc) to -diffuse large B-cell lymphoma
      * Burkitt Lymphoma
      * Lymphomatoid granulomatosis
   2. CD19+ indolent non-Hodgkin lymphoma including any of the following subtypes:

      * Follicular lymphoma (grade 1-3A)
      * Marginal zone lymphoma: Including splenic marginal zone lymphoma, nodal marginal zone lymphoma, and mucosa associated lymphoid tissue (MALT) lymphoma
      * Waldenstrom's Macrogloublinemia
      * Nodular lymphocyte predominant hodgkin lymphoma (with documented CD19 expression)
   3. Mantle cell Lymphoma
   4. Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Leukemia (SLL)
2. Prior Therapy Criteria Prior/Concurrent Therapy Related Criteria (dependent upon subtype - see below)

   1. Aggressive lymphoma: patients will qualify if any of the following scenarios are met below (radiation does not count as a line of therapy)

      * Relapse or persistent disease after ≥ 2 lines of systemic therapy OR
      * Refractory disease or relapse within 12 months of completion of 1st line systemic therapy OR
      * Refractory disease or relapse ≥ 1 line of therapy but not a candidate for autologous stem cell transplant
      * Patients with Burkitt lymphoma will qualify after ≥ 1 line of therapy regardless of the timing of relapse
   2. Indolent lymphoma:

      * Relapse or persistent disease after ≥ 2 lines of systemic therapy. (Neither single agent rituximab or radiation qualify as a line of therapy.)
   3. Mantle cell lymphoma:

      * Relapse or persistent disease after ≥ 1 line of systemic therapy. Neither single agent rituximab or radiation qualify as a line of therapy.
   4. Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma

      * Evidence of progression or intolerance after ≥ 2 lines of therapy. The following will qualify as a line of therapy for CLL/SLL:

        * systemic chemoimmunotherapy (e.g. BR, FCR, etc),
        * BTK inhibitor, BCL-2 inhibitor,
        * or PI3 Kinase inhibitor.
        * Neither single agent rituximab/obinutuzumab or radiation qualify as a line of therapy.
3. Clinical/Laboratory Criteria

   1. Participants must be at least 18 years old
   2. Participants must have a performance status of 0-2 on the ECOG scale
   3. Participants must have adequate caregiving support for CAR T-cell therapy as determined by the PI/Co-I.
   4. Participants must have measurable disease on cross section imaging by PET-CT and/or CT scans alone that is at least 1.5 cm in the longest diameter and measurable in two perpendicular dimensions as defined by IWG criteria. If participants with CLL do not have measurable disease on imaging, a bone marrow biopsy showing > 5% CLL involvement in the bone marrow will qualify for enrollment
   5. Participants that have received prior CD19 targeted therapy in the past they must have a tissue biopsy after completion of CD19 targeted therapy noting CD19 expression by either flowcytometry or immunohistochemistry (IHC). CD19 expression must be sufficient per PI/Co-I
   6. Adequate organ function

      * Bone marrow function as evidenced by the following (unless directly attributable to disease within the bone marrow) within 14 days prior to registration.

        * Platelet count ≥ 50,000 cells/mm3
        * ANC ≥ 750 cells/mm3
        * Absolute lymphocyte count ≥ 150 cells/ mm3
      * Hepatic function as evidenced by the following within 14 days prior to registration.

        * Serum bilirubin ≤ 1.5 X ULN unless attributed to Gilbert's syndrome or hemolysis or lymphoma involvement
      * Cardiac

        * No clinically significant ECG findings per PI/Co-I
      * Pulmonary

        * Oxygen saturation > 90% on room air
      * Renal function as evidenced by the following within 14 days prior to registration.

        * Serum creatinine ≤ 2 mg/dL or creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 60 mL/min
   7. Participants with hepatitis B virus infection must have undetectable viral load and on suppressive therapy within 14 days prior to registration and no evidence of HBV related hepatic damage.
   8. Participants with Hepatitis C infection must have complete eradication therapy completed, have no evidence of HCV related damage and have undetectable viral load within 14 days of registration.
   9. Participants with known human immunodeficiency virus (HIV)-infection must be receiving anti- retroviral therapy and have an undetectable viral load test within 14 days prior to registration.
   10. WOCBP should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below. FCBP must have negative serum or urine pregnancy within 7 days prior to registration.
   11. Men with female partners who are of childbearing potential: Recommendations for male and partner to use at least two effective contraceptive methods, as described above, during the study.
   12. Participants are able to understand and voluntarily sign consent prior to any study related assessments or procedures are performed.

Exclusion Criteria:

Participants eligible for study participation CANNOT meet any of the following criteria:

1. Prior/Concurrent Therapy Related Criteria Guidelines regarding when lymphoma directed therapy should be stopped prior to leukapheresis, lymphodepleting chemotherapy, and CAR T-cell infusion are detailed in the protocol. These criteria must be planned to be met for all patients.
2. Clinical/Laboratory Criteria

   1. Women who are pregnant or breast-feeding.
   2. Participants with active CNS lymphoma. Participants can have a history of active CNS lymphoma as outline in protocol
   3. Participants with evidence of Graft vs Host Disease from allogeneic stem cell transplant are ineligible unless it is either grade 1 involvement of the skin or not requiring systemic immunosuppression.
   4. Participants with uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
   5. Participants with a history of stroke or intracranial hemorrhage within 6 months prior to registration. Any CNS disorder that would serve as a major barrier in evaluating neurotoxicity/ICANS per enrolling physician
   6. Participants with prior history of malignancy other than lymphoma unless subject is free of disease for more than 1 year from signing consent. Exceptions include the following:

      * Basal cell carcinoma of the skin
      * Squamous cell carcinoma of the skin
      * Carcinoma in situ of the cervix or breast
      * Previously treated localized prostate cancer with normal PSA levels
   7. Participants with primary immunodeficiency or history of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 1 year.
   8. Participants with receipt of live vaccine within 28 days prior to registration.
   9. Participants with history of autologous stem cell transplant within the last 60 days or allogeneic stem cell transplant within the last 90 days or CAR T-cell therapy within the last 180 days.
   10. Participants with a history of severe immediate hypersensitivity reaction to any of the agents used in the study
   11. Participants with any other illness that in the opinion of the investigator, would exclude the patient from participating in this study.
   12. Participants must not have evidence of active CNS lymphoma involvement. This includes parenchymal, spinal cord, meningeal, or cerebrospinal fluid involvement. Patients with history of CNS involvement must have documented remission by contrast-enhanced MRI imaging and CSF evaluation for at least 60 days prior to registration.
   13. Patients must not have any unstable angina, or myocardial infarction within the last 6 months, or symptoms consistent with NYHA CHF classification III or IV
   14. Participants with receipt of live vaccine within 28 days prior to registration.
   15. Participants with history of autologous stem cell transplant within the last 60 days or allogeneic stem cell transplant within the last 90 days or CAR T-cell therapy within the last 180days.
   16. Participants with a history of severe immediate hypersensitivity reaction to any of the agents used in the study
   17. Participants with any other illness that in the opinion of the investigator, would exclude the patient from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
MTD/MAD/RP2D evaluation | 12 months
  Maximum tolerated dose (MTD), maximum administered dose (MAD) and the recommended phase 2 dose (RP2D) of CD19-CD34t metabolically programmed CAR T-cells
CRS occurrence evaluation | Duration of study, up to 24 months
  Rate of grade 3 or higher cytokine release syndrome(CRS)
ICANS occurrence evaluation | Duration of study, up to 24 months
  rate of grade 3 or higher immune effector cell-associated neurotoxicity syndrome (ICANS)

SECONDARY OUTCOMES:
Overall response and complete remission rate | 12 months
  1. Anti-tumor activity of CD19-CD34t metabolically programmed CAR T-cell therapy in adult patients with relapsed or refractory CD19 B-cell NHL or CLL/SLL based on overall response rate (ORR) and complete remission (CR) rate. The response rate for patients with NHL will be determined by the 2014 Lugano IWG criteria. The response rate for CLL/SLL patients will be determined by the 2018 iwCLL criteria
Progression free survival, duration of response, overall survival evaluations | 12 months
  Anti-tumor activity of CD19-CD34t metabolically programmed CAR T-cell therapy in adult patients with relapsed or refractory CD19 B-cell NHL or CLL/SLL based on progression free survival (PFS), duration of response (DOR), and overall survival (OS)
ORR and CR evaluation at the RP2D | Duration of study, up to 24 months
  Anti-tumor activity of CD19-CD34t metabolically programmed CAR T-cell therapy in adult patients with relapsed or refractory CD19 B-cell NHL or CLL/SLL treated at the RP2D based on ORR and CR rate. The response rate for patients with NHL will be determined by the 2014 Lugano IWG criteria. The response rate for CLL/SLL patients will be determined by the 2018 iwCLL criteria
PFS, DOR and OS evaluation at the RP2D | Duration of study, up to 24 months
  Anti-tumor activity of CD19-CD34t metabolically programmed CAR T-cell therapy in adult patients with relapsed or refractory CD19 B-cell NHL or CLL/SLL treated at the RP2D based on PFS, DOR and OS.
Safety evaluation at the RP2D | Duration of study, up to 24 months
  Safety of CD19-CD34t metabolically programmed CAR T-cells at the RP2D, including all grade incidence of CRS and ICANS

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hess, PHD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No